CLINICAL TRIAL: NCT01091259
Title: Phase II Study of Irinotecan in Combination With Bevacizumab for the Treatment of Recurrent Ovarian Cancer.
Brief Title: Irinotecan and Bevacizumab for Recurrent Ovarian Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NYU 09-0029
Record Dates: First submitted 2010-03-19; First posted 2010-03-23 (Estimated); Results first posted 2015-10-19 (Estimated); Last update posted 2015-11-24 (Estimated); Status verified 2015-10

CONDITIONS: Ovarian Cancer; Fallopian Tube Cancer; Primary Peritoneal Carcinoma
Keywords: antibody therapy; chemotherapy; biologic therapy; combination therapy
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms | interventions — Irinotecan; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Irinotecan with Bevacizumab (Experimental): Irinotecan is administered every 3 weeks at a dose of 175 mg/m^2, bevacizumab is administered at 15 mg/kg every 3 weeks. Irinotecan is administered before bevacizumab. Patients will continue on therapy until evidence of disease progression, or until development of adverse events that prevent further treatment, or if the patients wishes to discontinue therapy.
  Interventions: Drug: Irinotecan; Drug: Bevacizumab

INTERVENTIONS:
Drug: Irinotecan
  Other Names: Camptosar; CPT-11
Drug: Bevacizumab
  Other Names: Avastin

SUMMARY:
The purpose of the study is to evaluate the efficacy and toxicity of irinotecan in the treatment of women with recurrent epithelial ovarian cancer or primary peritoneal cancer when combined with bevacizumab.

DETAILED DESCRIPTION:
Accumulating data suggests that angiogenesis plays a critical role in the formation and development of a number of solid tumors including ovarian cancer. For women with ovarian cancer, a direct relationship between vascular endothelial growth factor (VEGF) expression and tumor vascularity has been documented. In vivo and in vitro data has demonstrated that increased angiogenesis and microvessel density are negative prognostic factors for women with ovarian cancer. These observations have fueled interest in incorporating anti-angiogenic agents into ovarian cancer treatment regimens.

Several phase II trials of irinotecan in patients with epithelial ovarian cancer showed that the drug had efficacy in both chemotherapy-naïve patients and in those who had been previously treated with standard therapies, including platinum-based compounds, radiation, or both. Combination of bevacizumab, an antibody against VEGF, and irinotecan was studied in colorectal cancer and malignant brain neoplasms. In these trials, the combination was shown to be safe and effective.

The purpose of this study is to evaluate the efficacy and toxicity of irinotecan in the treatment of women with recurrent epithelial ovarian cancer or primary peritoneal cancer when combined with bevacizumab. In this phase II open-label study patients will be treated with bevacizumab 15 mg/kg and irinotecan 175mg/m^2 every 3 weeks. Patients will undergo pre-treatment evaluation within 4 weeks of enrolling into the study. Clinical and laboratory evaluation will be performed every 3 weeks. Imaging studies and CA-125 measurements will be used to assess response to treatment.

ELIGIBILITY:
Inclusion Criteria:

* Women with recurrent epithelial ovarian cancer, fallopian tube cancer, or primary peritoneal carcinoma
* Patient should have measurable or evaluable disease as defined by the following.
* Measurable disease: At least one lesion that can be accurately measured in at least one dimension (longest dimension to be recorded). Each lesion must be ≥ 20 mm when measured by conventional techniques, including palpation, plain x-ray, CT and MRI, or ≥ 10 mm when measured by spiral CT.
* Evaluable (nonmeasurable) disease: Patients who do not meet measurable criteria will be eligible having known disease with CA125 levels >50 U/mL on two occasions at least one week apart. They will be considered for CA125 response criteria.
* Any number of prior chemotherapy regimens
* Any number of prior bevacizumab-containing regimens
* No chemotherapy within the last 2 weeks prior to initiating this study.
* Karnofsky Performance status score ≥ 60%.
* Patients must have a life expectancy ≥ 12 weeks.
* Patients must be at least 18 years of age.
* Patients must understand and willingly sign an approved informed consent.

Exclusion Criteria:

* Inability to comply with study and/or follow-up procedures
* Life expectancy of less than 12 weeks
* Current, recent (within 4 weeks of the first infusion of this study), or planned participation in an experimental drug study other than a Genentech-sponsored bevacizumab cancer study
* Active malignancy, other than superficial basal cell and superficial squamous (skin) cell, or carcinoma in situ of the cervix within last five years

Bevacizumab-Specific Exclusions

* Inadequately controlled hypertension (defined as systolic blood pressure > 150 mmHg and/or diastolic blood pressure > 100 mmHg)
* Prior history of hypertensive crisis or hypertensive encephalopathy
* New York Heart Association (NYHA) Grade II or greater congestive heart failure
* History of myocardial infarction or unstable angina within 6 months prior to Day 1
* History of stroke or transient ischemic attack within 6 months prior to Day 1 Known central nervous system disease, except for treated brain metastasis
* Treated brain metastases are defined as having no evidence of progression or hemorrhage after treatment and no ongoing requirement for dexamethasone, as ascertained by clinical examination and brain imaging (MRI or CT) during the screening period. Anticonvulsants (stable dose) are allowed. Treatment for brain metastases may include whole brain radiotherapy (WBRT), radiosurgery (RS; Gamma Knife, LINAC, or equivalent) or a combination as deemed appropriate by the treating physician. Patients with CNS metastases treated by neurosurgical resection or brain biopsy performed within 3 months prior to Day 1 will be excluded
* Significant vascular disease (e.g., aortic aneurysm, requiring surgical repair or recent peripheral arterial thrombosis) within 6 months prior to Day 1
* History of hemoptysis (>= 1/2 teaspoon of bright red blood per episode) within 1 month prior to Day 1
* Evidence of bleeding diathesis or significant coagulopathy (in the absence of therapeutic anticoagulation)
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to Day 1 or anticipation of need for major surgical procedure during the course of the study
* Core biopsy or other minor surgical procedure, excluding placement of a vascular access device, within 7 days prior to Day 1
* History of abdominal fistula or gastrointestinal perforation within 6 months prior to Day 1
* Serious, non-healing wound, active ulcer, or untreated bone fracture
* Proteinuria as demonstrated by a UPC ratio >= 1.0
* Known hypersensitivity to any component of bevacizumab
* Pregnancy (positive pregnancy test) or lactation. Use of effective means of contraception (men and women) in subjects of child-bearing potential
* History of abdominal fistula or intra-abdominal abscess within 6 months prior to start.
* Any history of prior gastrointestinal perforation
* Patients believed to possibly be at higher than average risk of perforation, including symptoms or findings of partial or complete bowel obstruction, history of fistula, patients requiring parenteral nutrition and hydration, and those with history of prior perforation due to tumor or perforation within last 6 months from other causes will be excluded from study
* Patients with evidence of abdominal free air not explained by paracentesis

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2010-03; Primary Completion 2014-02 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Franco Muggia, MD, Principal Investigator — New York Unviersity Cancer Institute
Locations (2):
- United States (2):
  - Bellevue Hospital Center (NYU Langone Medical Center affiliate), New York, New York
  - New York University Clinical Cancer Center, New York, New York

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From April 2010 to May 2013, 29 patients were enrolled from New York University Langone Medical Center.
Groups:
- Irinotecan With Bevacizumab: Irinotecan is administered every 3 weeks at a dose of 175 mg/m^2, bevacizumab is administered at 15 mg/kg every 3 weeks. Irinotecan is administered before bevacizumab. Patients will continue on therapy until evidence of disease progression, or until development of adverse events that prevent further treatment, or if the patients wishes to discontinue therapy.
  Irinotecan
  Bevacizumab
Period: Overall Study
Arm/Group | Irinotecan With Bevacizumab
Started | 29
Completed | 24 (Number of patients who had at least 2 cycles of treatments)
Not Completed | 5
Not completed — Adverse Event | 3
Not completed — Lack of Efficacy | 2

BASELINE CHARACTERISTICS:
Arm/Group | Irinotecan With Bevacizumab
Number analyzed (Participants) | 29
Age, Continuous [Median (Full Range); unit: years] | 62 [47 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 24
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 23
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 29
Number of prior regimens [Median (Full Range); unit: Regimens] | 5 [1 to 12]

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS) Rate at 6 Months
Description: The PFS rate at 6 months is the percentage of patients that experience a PFS event during the first 6 months in the study. The PFS is defined as the time from date of first dose of study medication to the date of first documented disease progression, or death from any cause, whichever is first. Patients who die without a reported prior progression will be considered to have progressed on the day of their death. Progression is evaluated by Response and Evaluation Criteria in Solid Tumor (RECIST) 1.0 or CA125 criteria if no measurable disease as doubling of CA125 levels from either the upper limit of normal or the nadir CA125 level.
Time Frame: 6 months from the start of treatment
Population: Intent-to-treat population.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Irinotecan With Bevacizumab
Number analyzed (Participants) | 29
percentage of patients | 55.2 [39.7 to 76.6]

2. Secondary Outcome: Overall Response Rate (ORR)
Description: ORR is defined as the percentage of all patients with confirmed partial response (PR) or complete response (CR). PR and CR are evaluated by RECIST 1.0 or CA125 if no measurable disease (PR: CA125 decreases by > 50%; CR: CA125 decreases to the normal range).
Time Frame: up to 3 years
Population: Intent-to-treat population
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Irinotecan With Bevacizumab
Number analyzed (Participants) | 29
percentage of patients | 27.6 [12.7 to 47.2]

3. Secondary Outcome: Median Progression Free Survival
Description: Defined as the length of time from the start of treatment that half of the patients are still alive and without disease progression. Progression is evaluated by RECIST 1.0 or CA125 if no measurable disease (PR: CA125 decreases by > 50%; CR: CA125 decreases to the normal range; progression is defined on the basis of a confirmed doubling of CA125 levels from either the upper limit of normal or the nadir CA125 level)
Time Frame: up to 3 years
Population: Intent-to-treat
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Irinotecan With Bevacizumab
Number analyzed (Participants) | 29
months | 6.8 [5.1 to 12.1]

4. Secondary Outcome: Median Overall Survival
Description: Defined as the length of time from the start of treatment that half of the patients are still alive.
Time Frame: up to 3 years
Population: Intent-to-treat
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Irinotecan With Bevacizumab
Number analyzed (Participants) | 29
months | 15.4 [11.9 to 20.4]

5. Secondary Outcome: Number of Patients Who Experienced Grade 3 and Higher Toxicities
Time Frame: up to 3 years
Population: Any patients who had at least one dose of treatment
Measure: Number; unit: participants
Arm/Group | Irinotecan With Bevacizumab
Number analyzed (Participants) | 29
participants
  Diarrhea | 5
  Fatigue | 3
  Pain | 3
  Hypertension | 2
  Nausea | 2
  Proteinuria | 2
  Vomiting | 2
  Febrile neutropenia | 1
  GI obstruction: colon | 1
  GI perforation | 1
  Leukopenia | 1

ADVERSE EVENTS:
Time Frame: The adverse events (AEs) are collected from the start of the treatment till 30 days off treatment.
Description: All AEs regardless of attribution are reported.
Arm/Group | Irinotecan With Bevacizumab
Serious Adverse Events (participants affected / at risk) | 9/29
Other Adverse Events (participants affected / at risk) | 29/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Irinotecan With Bevacizumab (N=29)
Pain: Abdomen NOS (Gastrointestinal disorders) | 2
Colitis (Gastrointestinal disorders) | 1
Obstruction, GI: Colon (Gastrointestinal disorders) | 1
Perforation, GI: Colon (Gastrointestinal disorders) | 1
Seizure (Nervous system disorders) | 1
Dehydration (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 3
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Hemorrhage, GI: Liver (Hepatobiliary disorders) | 1
Hypertension (Cardiac disorders) | 1
Leukocytes (total WBC) (Investigations) | 1
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 1
Vomiting (Gastrointestinal disorders) | 1
Renal/Genitourinary - Other: hydronephrosis (Renal and urinary disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Irinotecan With Bevacizumab (N=29)
Distension/bloating, abdominal (Gastrointestinal disorders) | 3
Pain: Abdomen NOS (Gastrointestinal disorders) | 7
Neuropathy: cranial: CN XI Motor-sternomastoid and trapezius (Nervous system disorders) | 1
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 2
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 2
Hair loss/alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 7
Anorexia (Gastrointestinal disorders) | 8
Mood alteration: Anxiety (Psychiatric disorders) | 1
Pain: Joint (Musculoskeletal and connective tissue disorders) | 3
AST, SGOT(serum glutamic oxaloacetic transaminase) (Investigations) | 3
Pain: Back (Musculoskeletal and connective tissue disorders) | 5
Creatinine (Metabolism and nutrition disorders) | 2
Pain: Bone (Musculoskeletal and connective tissue disorders) | 1
Pain: Breast (Reproductive system and breast disorders) | 2
Infection with normal ANC or Grade 1 or 2 neutrophils: Bronchus (Infections and infestations) | 1
Hemorrhage, GI: Colon (Gastrointestinal disorders) | 1
Constipation: (Gastrointestinal disorders) | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Dehydration (Gastrointestinal disorders) | 1
Mood alteration: Depression (Psychiatric disorders) | 3
Diarrhea (Gastrointestinal disorders) | 19
Dizziness (Nervous system disorders) | 1
Dry eye syndrome (Eye disorders) | 1
Dry mouth/salivary gland (xerostomia) (Gastrointestinal disorders) | 1
Taste alteration (dysgeusia) (Gastrointestinal disorders) | 3
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 5
Bruising (in absence of Grade 3 or 4 thrombocytopenia): (Skin and subcutaneous tissue disorders) | 1
Hemorrhage, pulmonary/upper respiratory: Nose (Respiratory, thoracic and mediastinal disorders) | 2
Rash: erythema multiforme (e.g., Stevens-Johnson syndrome, toxic epidermal necrolysis) (Skin and subcutaneous tissue disorders) | 1
Mood alteration: Euphoria (Psychiatric disorders) | 1
Pain: Face (General disorders) | 1
Fatigue (asthenia, lethargy, malaise) (General disorders) | 16
Flatulence (Gastrointestinal disorders) | 2
Flushing (Vascular disorders) | 2
Gastritis (including bile reflux gastritis) (Gastrointestinal disorders) | 2
Hematoma (Vascular disorders) | 1
Hemoglobin (Blood and lymphatic system disorders) | 7
Hemorrhoids (Gastrointestinal disorders) | 1
Pain: Head/headache (Nervous system disorders) | 9
Hiccoughs (hiccups, singultus) (Respiratory, thoracic and mediastinal disorders) | 1
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 3
Hypertension (Cardiac disorders) | 10
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 1
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 1
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 1
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 2
Hypothermia (General disorders) | 1
Flu-like syndrome (General disorders) | 1
Voice changes/dysarthria (e.g., hoarseness, loss or alteration in voice, laryngitis) (Respiratory, thoracic and mediastinal disorders) | 4
Leukocytes (total WBC) (Investigations) | 5
Rash: hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 1
Lymphopenia (Investigations) | 1
Memory impairment (Nervous system disorders) | 3
Muscle weakness, generalized or specific area (not due to neuropathy): Whole body/generalized (Musculoskeletal and connective tissue disorders) | 2
Pain: Muscle (Musculoskeletal and connective tissue disorders) | 3
Nausea (Gastrointestinal disorders) | 19
Pain: Neck (Musculoskeletal and connective tissue disorders) | 1
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 2
Pain: Extremity-limb (Musculoskeletal and connective tissue disorders) | 3
Pain: Pain NOS (General disorders) | 1
Pain: Pelvis (Reproductive system and breast disorders) | 3
Neuropathy: sensory (Nervous system disorders) | 3
Pain: Throat/pharynx/larynx (Respiratory, thoracic and mediastinal disorders) | 1
Platelets (Investigations) | 6
Hemorrhage, pulmonary/upper respiratory: Pleura (Respiratory, thoracic and mediastinal disorders) | 2
Infection with normal ANC or Grade 1 or 2 neutrophils: Lung (pneumonia) (Infections and infestations) | 1
Urinary frequency/urgency (Renal and urinary disorders) | 1
Proteinuria (Metabolism and nutrition disorders) | 3
INR (International Normalized Ratio of prothrombin time) (Investigations) | 1
Pruritus/itching (Skin and subcutaneous tissue disorders) | 2
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 3
Allergic rhinitis (including sneezing, nasal stuffiness, postnasal drip) (Respiratory, thoracic and mediastinal disorders) | 3
Rigors/chills (General disorders) | 1
Salivary gland changes/saliva (Gastrointestinal disorders) | 1
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 1
Infection with normal ANC or Grade 1 or 2 neutrophils: Skin (cellulitis) (Infections and infestations) | 2
Mucositis/stomatitis (functional/symptomatic): Oral cavity (Gastrointestinal disorders) | 4
Sweating (diaphoresis) (General disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 1
Dental: teeth (Gastrointestinal disorders) | 1
Pain: Dental/teeth/peridontal (Gastrointestinal disorders) | 4
Pain: Urethra (Renal and urinary disorders) | 4
Infection with normal ANC or Grade 1 or 2 neutrophils: Urinary tract NOS (Infections and infestations) | 1
Vaginal discharge (non-infectious) (Reproductive system and breast disorders) | 2
Vision-blurred vision (Eye disorders) | 1
Vomiting (Gastrointestinal disorders) | 16
Weight loss (General disorders) | 4
Alkaline phosphatase (Investigations) | 2
Allergic reaction (Immune system disorders) | 1
Gastrointestinal- Other: increased salivation (Gastrointestinal disorders) | 2
Dermatology/Skin - Other: skin sensitivity (Skin and subcutaneous tissue disorders) | 1
Hemorrhage, GI: oral cavity (Gastrointestinal disorders) | 1
Infection - Other: Peritoneal Herpes Simplex (Infections and infestations) | 1
Musculoskeletal/Soft Tissue - Other: cramping hands (Musculoskeletal and connective tissue disorders) | 1
Ocular/Visual - Other: visual changes (Eye disorders) | 1
Pain: rectum (Gastrointestinal disorders) | 1
Nasal cavity//paranasal sinus reactions (Respiratory, thoracic and mediastinal disorders) | 1
Edema: limb (General disorders) | 2
Hemorrhage, pulmonary/upper respiratory: nose (Respiratory, thoracic and mediastinal disorders) | 1
Infection with unknown ANC: UTI (Infections and infestations) | 1
Pain: sinus (Respiratory, thoracic and mediastinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes